CLINICAL TRIAL: NCT03430999
Title: SUNCIST: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Ascending, Single-Dose Study to Assess the Safety, Tolerability, Pharmacokinetics of Intravenous Administration of Calmangafodipir in Healthy Japanese and Caucasian Subjects
Brief Title: SUNCIST: A Study of Calmangafodipir in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egetis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PP06466
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)
MeSH Terms: interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Japanese) Calmangafodipir (Experimental)
  Interventions: Drug: Calmangafodipir
- Group 1 (Japanese) Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Group 2 (Caucasian) Calmangafodipir (Experimental)
  Interventions: Drug: Calmangafodipir
- Group 2 (Caucasian) Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calmangafodipir — Single ascending doses of 2 μmol/kg, 5 μmol/kg, and 10 μmol/kg
  Arms: Group 1 (Japanese) Calmangafodipir; Group 2 (Caucasian) Calmangafodipir
Drug: Placebo — Placebo
  Arms: Group 1 (Japanese) Placebo; Group 2 (Caucasian) Placebo

SUMMARY:
Randomized, double-bline, placebo-controlled, single dose study comparing the pharmacokinetics (PK) and safety of PP095-01 in Japanese and non-Asian (eg, Caucasian) subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI within 18.0 to 30.0 kg/m2 and body weight not less than 50 kg
* Blood pressure between 90 and 140 mmHg systolic, and no higher than 90 mmHg diastolic
* Non-smoker or not smoking for at least 12 months
* Be first generation Japanese (For Group 1 only), defined as:

  1. Born in Japan
  2. Has 2 Japanese biological parents and 4 Japanese biological grandparents
  3. Has lived outside of Japan for less than 5 years
  4. Has made no significant changes in lifestyle, including diet, since leaving Japan

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry, urinalysis, physical exam, vital signs, or electrocardiogram at screening
* Has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV; has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening.
* Has a history of drug or alcohol abuse
* Has previously received calmangafodipir or mangafodipir
* Welders, mine workers, or other workers in occupations (current or past) where high manganese exposure is likely

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | From signing of informed consent through the last follow up visit (up to Day 10)
  Subject incidence of treatment-emergent adverse events (TEAEs), which may include changes in laboratory safety tests, electrocardiograms (ECG), and vital signs.

SECONDARY OUTCOMES:
Cmax | predose and 1 min, 15 min, 30 min, 1 hour, 4 hours, and 8 hours postdose
  Maximum plasma concentration during a dosing interval
tmax | predose and 1 min, 15 min, 30 min, 1 hour, 4 hours, and 8 hours postdose
  Time to reach maximum plasma concentration
AUC(0-last) | predose and 1 min, 15 min, 30 min, 1 hour, 4 hours, and 8 hours postdose
  Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration
Ae | 4 hours post-dose and 24 hours post-dose
  Amount of manganese and zinc excreted into urine
Ae% | 4 hours and 24 hours post-dose
  Percent of study drug manganese excreted into urine

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No